CLINICAL TRIAL: NCT04673019
Title: Nurse AMIE for Echo Show: Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other); American Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00016221
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a partial crossover trial in which immediate treatment group participants receive the Nurse AMIE intervention in full for 3 months, then continue Nurse AMIE (without navigation) for 3 months, while the delayed intervention group will not receive an intervention for 3 months, followed by receiving the Nurse AMIE full intervention with navigation for 3 months. The primary comparisons will be between the immediate treatment and delayed treatment groups over the first 3 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): The immediate intervention group will receive the intervention at the time of consent (baseline) and will be enrolled in the intervention for a total of 6 months:
  * Months 1- 3 (Approximately Day 1-Day 90)
    * Participant will receive the Echo Show, a pedometer (to track their steps) and an exercise band (to complete the exercise interventions).
    * Use of Nurse AMIE while receiving intervention phone calls from a study facilitator. We are interested in learning whether the phone calls are necessary or if the Nurse AMIE platform can stand alone and see the same effect.
  * Months 4-6 (Approximately Day 91-180) o Participant will continue to use Nurse AMIE, but without phone calls from study facilitator
  Interventions: Behavioral: Nurse AMIE (Addressing Metastatic Individuals Every day)
- Delayed Intervention (Other): The delayed intervention group will receive the intervention 3 months after consent (3 months of no intervention followed by with 3 months of intervention, for a total of 6 months); the participant will follow the pattern listed below:
  * Months 1- 3 Approximately (Day 1-Day 90)
    o No use of Nurse AMIE
  * Months 4-6 (Approximately Day 91-180)
    * Participant will receive the Echo Show, a pedometer (to track their steps) and an exercise band (to complete the exercise interventions).
    * Use of Nurse AMIE while receiving intervention phone calls from a study facilitator
  Interventions: Behavioral: Nurse AMIE (Addressing Metastatic Individuals Every day)

INTERVENTIONS:
Behavioral: Nurse AMIE (Addressing Metastatic Individuals Every day) — Supportive Care Platform (behavioral interventions that are offered based on answers to daily symptom rating questions). Interventions offered include walking, balance, strength exercise, guided relaxation, CBT, DBT, soothing music.

SUMMARY:
The Nurse AMIE platform has been modified for use as an Amazon Alexa skill for use on the Echo Show device. The investigators will recruit women receiving treatment for metastatic breast cancer and randomize patients to receive standard treatment (control) or the Nurse AMIE for Echo Show program. Nurse AMIE is a supportive care program for women undergoing chemotherapy and helps manage symptoms. The investigators will test the feasibility of using the Nurse AMIE program as well as its effectiveness at managing symptoms.

DETAILED DESCRIPTION:
The investigators will recruit 42 MBC patients and randomize them into a partial crossover trial in which immediate treatment group participants receive the Nurse AMIE intervention in full for 3 months, then continue Nurse AMIE (without navigation) for 3 months, while the delayed intervention group will not receive an intervention for 3 months, followed by receiving the Nurse AMIE full intervention with navigation for 3 months. The primary comparisons will be between the immediate treatment and delayed treatment groups over the first 3 months.

Intervention. Participants will all receive an Amazon Echo Show device, WiFi connection (if patients do not already have one), pedometer, and resistance bands. Each day, the participant will open the Nurse AMIE for Echo Show, which will result in the daily greeting. After the greeting, participants will be asked to provide a verbal rating of their symptoms (e.g., pain, sleep, fatigue, and distress).

After completing the symptom survey, Nurse AMIE will use an algorithm to discern which of the intervention modules to offer as assistance for the reported symptoms. These interventions include exercise, guided relaxation, cognitive behavioral therapy, and soothing music. These guideline-based interventions are provided as audio files or YouTube-style videos. In addition, Nurse AMIE provides a daily educational nutrition tip as well as recipes designed to be of interest to people undergoing chemotherapy.

Each week, the participant will receive a phone call from the study navigator. This navigator will monitor symptom ratings daily and will discuss symptoms, interventions, and step goals with the participant each week.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with metastatic breast cancer receiving care at PSCI
2. Age: ≥18years of age
3. Personal in-home Wi-Fi access
4. Personal device capable of receiving telephone calls for weekly study facilitator check-ins
5. Fluent in written and spoken English
6. Sufficient vision/hearing to use the Alexa Echo Show.

Exclusion Criteria:

1. ECOG Performance Status score of >2
2. Patients with significant medical or psychiatric conditions (beyond breast cancer, its treatment, and its symptoms) that in the opinion of the research team exclude the subject from participation.
3. Receiving any behavioral intervention.
4. Pregnant
5. Cognitive impairment
6. Life expectancy of less than 6 months as determined by the treating physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - the proportion of patients who interact with the tablet for at least one month | 90 days
  The proportion of women who consent, take a tablet home, who actually interact with the Nurse AMIE platform at least 30 out of 90 possible days
Acceptability - the proportion of patients who agree to participate | baseline
  The proportion of women who agree to participate among those deemed eligible and cleared by oncologist.

SECONDARY OUTCOMES:
Physical Function: Short Physical Performance Battery (SPPB) | baseline
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Physical Function: Short Physical Performance Battery (SPPB) | month 3
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Physical Function: Short Physical Performance Battery (SPPB) | month 6
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Health-Related Quality of Life measured using the 36-Item Short Form Health Survey (SF-36) | baseline
  The SF-36 measures quality of life in the following domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well being, social functioning, pain, and general health. All items are scored from 0 to 100, with 100 being the highest level of functioning possible. Items are averaged to give ratings on each of 8 dimensions.
Health-Related Quality of Life measured using the 36-Item Short Form Health Survey (SF-36) | month 3
  The SF-36 measures quality of life in the following domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well being, social functioning, pain, and general health. All items are scored from 0 to 100, with 100 being the highest level of functioning possible. Items are averaged to give ratings on each of 8 dimensions.
Health-Related Quality of Life measured using the 36-Item Short Form Health Survey (SF-36) | month 6
  The SF-36 measures quality of life in the following domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well being, social functioning, pain, and general health. All items are scored from 0 to 100, with 100 being the highest level of functioning possible. Items are averaged to give ratings on each of 8 dimensions.
Sleep Quality and Sleep Problems | baseline
  measured using the Pittsburgh Sleep Quality Inventory. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Sleep Quality and Sleep Problems | month 3
  measured using the Pittsburgh Sleep Quality Inventory. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Sleep Quality and Sleep Problems | month 6
  measured using the Pittsburgh Sleep Quality Inventory. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Well-being measured using the Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B+4) | baseline
  This measure is specific to patients with breast cancer and measures well-being in several domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The items are rated from 0 to 4, and total scores for each domain are the sums of the items (0 being low well-being). The total FACT-B score is the sum of the domains, with scores ranging from 0 to 148, with 148 being the highest level of well-being possible.
Well-being measured using the Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B+4) | month 3
  This measure is specific to patients with breast cancer and measures well-being in several domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The items are rated from 0 to 4, and total scores for each domain are the sums of the items (0 being low well-being). The total FACT-B score is the sum of the domains, with scores ranging from 0 to 148, with 148 being the highest level of well-being possible.
Well-being measured using the Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B+4) | month 6
  This measure is specific to patients with breast cancer and measures well-being in several domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The items are rated from 0 to 4, and total scores for each domain are the sums of the items (0 being low well-being). The total FACT-B score is the sum of the domains, with scores ranging from 0 to 148, with 148 being the highest level of well-being possible.
Distress measured using the Penn State Cancer Institute Distress Inventory | baseline
  The PSCI Distress Inventory is a 5-item questionnaire, which measures distress associated with: practical problems, family problems, emotional problems, spiritual religious concerns, and physical problems. The responses are rated from 0 (no distress) to 10 (severe distress).
Distress measured using the Penn State Cancer Institute Distress Inventory | month 3
  The PSCI Distress Inventory is a 5-item questionnaire, which measures distress associated with: practical problems, family problems, emotional problems, spiritual religious concerns, and physical problems. The responses are rated from 0 (no distress) to 10 (severe distress).
Distress measured using the Penn State Cancer Institute Distress Inventory | month 6
  The PSCI Distress Inventory is a 5-item questionnaire, which measures distress associated with: practical problems, family problems, emotional problems, spiritual religious concerns, and physical problems. The responses are rated from 0 (no distress) to 10 (severe distress).
Pain Severity and Pain Interference measured by the Brief Pain Inventory (BPI) | baseline
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Pain Severity and Pain Interference measured by the Brief Pain Inventory (BPI) | month 3
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Pain Severity and Pain Interference measured by the Brief Pain Inventory (BPI) | month 6
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Fatigue measured using the Brief Fatigue Inventory (BFI) | baseline
  The BFI is a nine-item measure, with scores ranging from 0 being best/no fatigue, and 10 being fatigue as bad as imaginable. A global fatigue score is calculated as an average of the nine items.
Fatigue measured using the Brief Fatigue Inventory (BFI) | month 3
  The BFI is a nine-item measure, with scores ranging from 0 being best/no fatigue, and 10 being fatigue as bad as imaginable. A global fatigue score is calculated as an average of the nine items.
Fatigue measured using the Brief Fatigue Inventory (BFI) | month 6
  The BFI is a nine-item measure, with scores ranging from 0 being best/no fatigue, and 10 being fatigue as bad as imaginable. A global fatigue score is calculated as an average of the nine items.

OTHER OUTCOMES:
Physical Activity | Daily for 90 days
  measured using step counts recorded with an analog pedometer, self-reported to the Nurse AMIE platform by the participant each day
Usability as measured by the System Usability Scale (SUS) | month 3
  Ease of use of the Nurse AMIE for Echo Show platform will be assessed using the System Usability Scale (SUS). Each of the 10 items on this scale are rated from 0 to 4. Items are summed and multiplied by 2.5 to obtain the overall value of the usability. SUS scores range from 0 to 100, with the higher score indicating better ease of use.
Usability as measured by the System Usability Scale (SUS) | month 6
  Ease of use of the Nurse AMIE for Echo Show platform will be assessed using the System Usability Scale (SUS). Each of the 10 items on this scale are rated from 0 to 4. Items are summed and multiplied by 2.5 to obtain the overall value of the usability. SUS scores range from 0 to 100, with the higher score indicating better ease of use.
App Quality measured by the Mobile Application Rating Scale (U-MARS) | month 3
  Ease of use of the Nurse AMIE for Echo Show platform measured by the Mobile Application Rating Scale (U-MARS). Each item is rated from 1 (inadequate) to 5 (excellent). Items are summed to give subscores of Engagement, Functionality, Aesthetics, Information. These subscores can be averaged to give an app quality score. Further, there are two additional scores, the subjective quality and app-specific scores that are used to assess the participant's view of the quality of the app and the impact of the app on knowledge, attitudes, intentions, and change in target health behavior, respectively. The higher the score, the more favorable the app quality is.
App Quality measured by the Mobile Application Rating Scale (U-MARS) | month 6
  Ease of use of the Nurse AMIE for Echo Show platform measured by the Mobile Application Rating Scale (U-MARS). Each item is rated from 1 (inadequate) to 5 (excellent). Items are summed to give subscores of Engagement, Functionality, Aesthetics, Information. These subscores can be averaged to give an app quality score. Further, there are two additional scores, the subjective quality and app-specific scores that are used to assess the participant's view of the quality of the app and the impact of the app on knowledge, attitudes, intentions, and change in target health behavior, respectively. The higher the score, the more favorable the app quality is.
Comprehensive Symptom Assessment measured with the Patient-Generated Subjective Global Assessment (PG-SGA) | Weekly over a 3 month (90 day) intervention period
  The PG-SGA is a self-report assessment of symptoms related to cancer and its treatment. This checklist allows clinical care teams to understand the symptom burden that a participant is experiencing. Symptoms are assigned values with low values (e.g., 0) being the lowest symptom burden (favorable).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn H Schmitz, PhD, Principal Investigator — Penn State Milton Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Schmitz KH, Kanski B, Gordon B, Caru M, Vasakar M, Truica CI, Wang M, Doerksen S, Lorenzo A, Winkels R, Qiu L, Abdullah S. Technology-based supportive care for metastatic breast cancer patients. Support Care Cancer. 2023 Jun 20;31(7):401. doi: 10.1007/s00520-023-07884-3. PMID 37338627
- [Derived] Gordon BR, Qiu L, Doerksen SE, Kanski B, Lorenzo A, Truica CI, Vasekar M, Wang M, Winkels RM, Abdullah S, Schmitz KH. Addressing metastatic individuals everyday: Rationale and design of the nurse AMIE for Amazon Echo Show trial among metastatic breast cancer patients. Contemp Clin Trials Commun. 2023 Jan 16;32:101058. doi: 10.1016/j.conctc.2023.101058. eCollection 2023 Apr. PMID 36698743